CLINICAL TRIAL: NCT00928304
Title: An Open-Label, Non-Randomized Study to Evaluate the Efficacy and Safety of BAY94-9172 (ZK 6013443) Positron Emission Tomography (PET) for Detection of Cerebral ß-Amyloid in Individuals With Down Syndrome Compared to Individuals Without Down Syndrome
Brief Title: Phase II Study of Florbetaben (BAY94-9172) PET Imaging for Detection/Exclusion of Cerebral β-amyloid.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14311
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Down Syndrome; Amyloid Beta-protein
Keywords: Amyloid beta-protein; Down Syndrome
MeSH Terms: conditions — Down Syndrome; Plaque, Amyloid | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Florbetaben (BAY94-9172) (Experimental)
  Interventions: Drug: Florbetaben (BAY94-9172)

INTERVENTIONS:
Drug: Florbetaben (BAY94-9172) — 300 megabecquerels (MBq) as single IV injection of 2 to 10 mL

SUMMARY:
To determine the sensitivity of the visual assessment of BAY94-9172 PET images in detecting cerebral β-amyloid in individuals with Down Syndrome (DS) and specificity in individuals without DS. Given that individuals with Down Syndrome develop β-amyloid pathology over the age of 40, the clinical diagnosis of Down Syndrome will serve as the standard of truth.

ELIGIBILITY:
Inclusion Criteria:

Study participants were individuals with DS and healthy volunteers (HVs).

* Main inclusion criteria for individuals without DS

  * >=21 and <= 40 years of age
  * Mini-Mental State Examination (MMSE) >= 28
  * Clinical Dementia Rating (CDR) of 0
* Main inclusion criteria for individuals with DS

  * >= 40 years of age

Exclusion Criteria:

* Main exclusion criteria for both groups

  * Unstable medical or psychiatric condition, study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Sun City, Arizona
  - New Haven, Connecticut

REFERENCES:
- [Derived] Bullich S, Roe-Vellve N, Marquie M, Landau SM, Barthel H, Villemagne VL, Sanabria A, Tartari JP, Sotolongo-Grau O, Dore V, Koglin N, Muller A, Perrotin A, Jovalekic A, De Santi S, Tarraga L, Stephens AW, Rowe CC, Sabri O, Seibyl JP, Boada M. Early detection of amyloid load using 18F-florbetaben PET. Alzheimers Res Ther. 2021 Mar 27;13(1):67. doi: 10.1186/s13195-021-00807-6. PMID 33773598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two sites in the US.
Pre-assignment Details: A total of 130 subjects were screened. 21 subjects were considered as screen failures and were not enrolled into the study. 9 subjects did not meet the inclusion/exclusion criteria. 10 subjects withdrew their consent. 1 subject was lost to follow-up and 1 subjected exceeded the weight limit for the camera.
Groups:
- Down Syndrome Group: 39 Down Syndrome subjects received Florbetaben (BAY94-9172) : 300 megabecquerels (MBq) single IV injection of 2 to 10 mL
- Healthy Volunteer Group: 70 healthy volunteer subjects received Florbetaben (BAY94-9172): 300 MBq single IV injection of 2 to 10 mL
Period: Overall Study
Arm/Group | Down Syndrome Group | Healthy Volunteer Group
Started | 39 | 70
Completed | 39 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Down Syndrome subjects and healthy volunteers enrolled into the study were included in the Baseline Analysis Population
Groups:
- Subjects Enrolled in Study: All Down Syndrome and healthy volunteer subjects
Arm/Group | Subjects Enrolled in Study
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Down Syndrome Group | 46.3 (4.7)
  Healthy Volunteer Group | 27.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the Independent Visual Assessment of Detecting Cerebral Amyloid-beta in Individuals With Down Syndrome and Specificity in Subjects Without Down Syndrome
Description: The primary variables are sensitivity (percentage of DS subjects positive for cerebral beta-amyloid) and specificity (percentage of healthy volunteers negative for cerebral beta-amyloid) of brain uptake of florbetaben based on the majority read of the visual assessment by three independent blinded readers of PET images obtained 100 to 120 minutes post-injection of florbetaben.
Time Frame: 100-120 min
Population: All subjects in the down syndrome population and healthy volunteers were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Majority Read: Majority read of the visual assessment made by 3 independent readers of PET images from all subjects.
Arm/Group | Majority Read
Number analyzed (Participants) | 109
percentage of subjects
  Sensitivity | 46.15 [30.51 to 61.80]
  Specificity | 100.00 [100.00 to 100.00]

2. Secondary Outcome: Sensitivity Results in the Down Syndrome Age Subgroups
Description: The majority read sensitivity (percentage of DS subjects positive for cerebral beta-amyloid by majority read) was computed for the group of DS subjects with age equal to or below the median age (DS-young) and for DS subjects with age above the median age (DS-old). The median age was 46 yrs, with 3 subjects being exactly 46 yrs old. As defined, these subjects were assigned to the DS-young group.
Time Frame: 100 - 120 min
Population: All Down Syndrome subjects (n=39) were analyzed for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Majority Read (DS-Young): Majority Read results for Down Syndrome subjects with age <= 46 yrs
- Majority Read (DS-Old): Majority Read results for Down Syndrome subjects with age >46 yrs
Arm/Group | Majority Read (DS-Young) | Majority Read (DS-Old)
Number analyzed (Participants) | 21 | 18
percentage of subjects | 23.81 [5.59 to 42.03] | 72.22 [51.53 to 92.91]

3. Secondary Outcome: Quantitative Parameters Standard Uptake Value Ratio
Description: The Standard Uptake Value Ratios for florbetaben signal in the frontal cortex, posterior cingulate, lateral temporal cortex, parietal cortex, and cerebellum (white matter) were determined as a quantitative measure of tracer uptake. The SUV is defined as the ratio of (1) the tissue radioactivity concentration c (in MBq/kg) at time point t, and (2) the injected activity (in MBq, extrapolated to the same time t) divided by the body weight (in kg). These SUV numbers from regions of interest were then used to derive SUV ratios (SUVR) using the SUV from the cerebellar cortex as reference.
Time Frame: 100 - 120 min p.i.
Population: All Down Syndrome subjects and healthy volunteers enrolled in the study were included in this analysis
Measure: Mean (Standard Deviation); unit: SUVR
Groups:
- Down Syndrome Group: Subjects with Down Syndrome enrolled in the study
- Healthy Volunteer Group: Healthy volunteers enrolled in the study
Arm/Group | Down Syndrome Group | Healthy Volunteer Group
Number analyzed (Participants) | 39 | 70
SUVR
  frontal cortex | 1.396 (0.2488) | 1.146 (0.0749)
  posterior cingulate | 1.525 (0.2549) | 1.329 (0.1118)
  lateral temporal cortex | 1.350 (0.2265) | 1.132 (0.0623)
  parietal cortex | 1.391 (0.2594) | 1.138 (0.0742)
  cerebellum, white matter | 1.730 (0.2115) | 1.769 (0.1302)

4. Secondary Outcome: Consistency Between Visual and Quantitative Efficacy
Description: For a comparison of the results of the visual assessment with the quantitative assessment, descriptive Standardized Uptake Value Ratio (SUVR) statistics were computed separately for DS subjects with an abnormal/normal majority read of the PET scan (DS-PET+/DS-PET-). The SUV is defined as the ratio of (1) the tissue radioactivity concentration c (in MBq/kg) at time point t, and (2) the injected activity (in MBq, extrapolated to the same time t) divided by the body weight (in kg). These SUV numbers from regions of interest were then used to derive SUV ratios (SUVR) using the SUV from the cerebellar cortex as reference.
Time Frame: 100 - 120 min
Measure: Mean (Standard Deviation); unit: SUVR
Groups:
- Down Syndrome PET-positive (Majority Read): Down Syndrome subjects positive for cerebral beta-amyloid as determined by majority read
- Down Syndrome PET-negative (Majority Read): Down Syndrome subjects negative for cerebral beta-amyloid as determined by majority read
- Healthy Volunteer Group: All healthy volunteers enrolled in the study
Arm/Group | Down Syndrome PET-positive (Majority Read) | Down Syndrome PET-negative (Majority Read) | Healthy Volunteer Group
Number analyzed (Participants) | 18 | 21 | 70
SUVR
  frontal cortex | 1.566 (0.2372) | 1.249 (0.1451) | 1.146 (0.0749)
  posterior cingulate | 1.626 (0.2372) | 1.438 (0.2421) | 1.329 (0.1118)
  lateral temporal cortex | 1.498 (0.2396) | 1.223 (0.1092) | 1.132 (0.0623)
  parietal cortex | 1.557 (0.2567) | 1.250 (0.1620) | 1.138 (0.0742)
  cerebellum, white matter | 1.698 (0.2396) | 1.758 (0.1856) | 1.769 (0.1302)

ADVERSE EVENTS:
Time Frame: 8 days
Description: Adverse event data were collected from Day 1 (baseline) until Day 8 (secondary follow-up visit)
Groups:
- Down Syndrome Group: 39 Down Syndrome subjects received Florbetaben (BAY94-9172): 300 MBq single IV injection of 2 to 10 mL
Arm/Group | Down Syndrome Group | Healthy Volunteer Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/70
Other Adverse Events (participants affected / at risk) | 2/39 | 5/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Down Syndrome Group (N=39) | Healthy Volunteer Group (N=70)
Injection site hematoma (General disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less